Consent Form Version 2: 17<sup>th</sup> September 2020 IRAS Number: 286383





IRAS ID: 286383

Study Number:

Participant Identification Number for this trial:

## **CONSENT FORM**

Title of Project: Brain activity response to cues during gait in Parkinson's

Name of Researcher:

| Please initial the boxes that apply to you | Consent | |
|---|---|---|
| | (initial) | |
| I confirm that I have read and understand the information sheet dated (version) for the above study. I have had the opportunity to consider the information, ask questions and have had these answered satisfactorily. | | |
| I understand that my participation is voluntary and that I am free to withdraw at any time without giving any reason, without my medical care or legal rights being affected. | | |
| I consent to my GP being informed of my participation in this study. | | |
| I understand that relevant sections of my medical notes and data collected during the study may be looked at by individuals from the Sponsor and the NHS Trust, where it is relevant to my taking part in this research. I give permission for these individuals to have access to my records. | | |
| I give permission for my records / data to be used for this study. | | |
| I understand that my personal data (e.g. name, address) will be stored at Northumbria University within secure facilities for 12 months, after which it will be disposed of. | | |
| I understand that all of my study data will anonymised and stored at Northumbria University within secure facilities for 10 years, after which it will be disposed of. | | |
| I understand that all records are confidential and anonymous, and kept in locked filing cabinets which are accessed only by research staff working on this project. | | |
| I agree to participate in this study. | | |
| Additional (Optional items): | Consent | Decline |
| | (initial) | (initial) |
| I understand that the video and/or photographs will be stored on a secure computer under a participant study code (e.g. PD01) in the Clinical Gait laboratory, Northumbria University and will only leave the unit for the | | |

Consent Form Version 2: 17<sup>th</sup> September 2020 IRAS Number: 286383





| purposes agreed to below. I understand that my name and personal details |
|---|
| will not be kept with the video and, as such, I cannot be identified from it. |
| I consent to my facial features being recognisable on video / photography. |
| I consent to the use of video / photographs collected on the study for |
| internal staff training |
| • inclusion in presentations at national and international educational |
| meetings |
| inclusion in publications including academic journals and their |
| internet sites |
| I agree to be contacted about ethically approved research studies for |
| which I may be suitable. I understand that agreeing to be contacted does |
| not oblige me to participate in any further studies. |
| I agree for my anonymised data to be archived in a suitable discipline data |
| repository, and anonymised data may be used in future by other |
| researchers. |

Title of Project: Brain activity response to cues during gait in Parkinson's

| Signed | |
|------------------------|-------------|
| Printed Name | Date |
| Person taking consent: | |
| Printed name | Signed |
| Date | Designation |

Participant: